CLINICAL TRIAL: NCT00400543
Title: Effects of Continuous Positive Airway Pressure (CPAP) on Early Signs of Atherosclerosis in Patients With Obstructive Sleep Apnea: a Randomized Study
Brief Title: Early Signs of Atherosclerosis in Obstructive Sleep Apnea: Effects of Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SDC 2431/04/051
Record Dates: First submitted 2006-11-16; First posted 2006-11-17 (Estimated); Last update posted 2006-11-17 (Estimated); Status verified 2006-11

CONDITIONS: Obstructive Sleep Apnea; Atherosclerosis
Keywords: obstructive sleep apnea; arterial stiffness; atherosclerosis; CPAP; heart disease
MeSH Terms: conditions — Sleep Apnea, Obstructive; Atherosclerosis; Heart Diseases | interventions — Continuous Positive Airway Pressure

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP)

SUMMARY:
Obstructive sleep apnea (OSA) is associated with adverse cardiovascular outcomes, including acute myocardial infarction and stroke. Atherosclerosis is an important step for these events. Recent studies demonstrated the independent association between OSA and validated markers of atherosclerosis. However, the impact of treatment with continuous positive airway pressure (CPAP) on these markers is unknown.

The purpose of this study is to determine whether CPAP therapy can reverses early signs of atherosclerosis in apparently healthy OSA patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is characterized by recurrent episodes of partial or complete obstruction of the upper airway during sleep resulting in oxygen desaturation and arousals from sleep. OSA is recognized as an important public health problem, affecting 9 and 24 % of middle-aged females and males, respectively. There is now compelling evidence that severe OSA is associated with increased cardiovascular morbidity and mortality, mainly due to acute myocardial infarction and stroke. Moreover, the current standard treatment with application of continuous positive airway pressure (CPAP) during the night was associated with decreased non-fatal and fatal cardiovascular events.

There are several mechanisms associated with OSA that are potentially harmful to the cardiovascular system, including sympathetic activation, systemic inflammation, production of reactive oxygen species, and endothelial dysfunction. Together, all these factors could contribute to atherosclerosis progression, a key mechanism involved in the genesis of myocardial infarction and stroke. For instance, we recently described the presence of early signs of atherosclerosis in otherwise healthy OSA subjects as characterized by alterations in validated markers of atherosclerosis, including increased arterial stiffness, evaluated by pulse wave velocity (PWV), as well as intima-media thickness (IMT) and carotid diameter (CD). All theses vascular abnormalities correlated significantly with the severity of the OSA.

In this study, we will perform a randomized study to evaluate the impact of CPAP therapy on PWV, IMT and CD as well as in catecholamine and C reactive protein. We made the hypothesis that CPAP promotes beneficial effects on atherosclerosis, independent of the other factors, such as blood pressure and cholesterol levels. To this end, we only will study young OSA patients that were free of co-morbidities. Patients will be randomized to no treatment (Control) or CPAP for 4 months. Evalutations will be performed at baseline and after 4 months.

ELIGIBILITY:
Inclusion Criteria:

* Males with recent sleep study (<1 month) showing severe obstructive sleep apnea, defined as at least 30 events of apnea and hypopnea per hour of sleep.

Exclusion Criteria:

* Age >60 years old, body mass index (BMI) >35 kg/m2, diabetes mellitus, hypertension, cerebrovascular, aortic, heart, and valvar heart diseases, renal failure, arrhythmias, smoking habit, and chronic use of medications, including statins.

Ages: 30 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24
Dates: Start 2004-01; Study Completion 2006-07

PRIMARY OUTCOMES:
Arterial stiffness (evaluated by PWV)
Intima media thickness (IMT)
Carotid diameter (CD)

SECONDARY OUTCOMES:
24h blood pressure monitoring
plasma catecholamine
C-reactive protein (CRP)

CONTACTS AND LOCATIONS:
Overall Officials: Luciano F Drager, MD, Principal Investigator — InCor Heart Institute
Locations (1):
- Heart Institute (InCor) - University of São Paulo Medical School, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Drager LF, Bortolotto LA, Figueiredo AC, Krieger EM, Lorenzi GF. Effects of continuous positive airway pressure on early signs of atherosclerosis in obstructive sleep apnea. Am J Respir Crit Care Med. 2007 Oct 1;176(7):706-12. doi: 10.1164/rccm.200703-500OC. Epub 2007 Jun 7. PMID 17556718